CLINICAL TRIAL: NCT00298376
Title: Oral Tolerance in Cow's Milk Allergy in the Infant: Role of CD4+CD25+ T Cells and Intestinal Microflora
Brief Title: Oral Tolerance in Cow's Milk Allergy in the Infant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Other Study IDs: 2005.389
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Cow's Milk Allergy
Keywords: Cow's milk allergy,; food allergy; oral tolerance,; infant,; regulatory T cells,; intestinal microflora
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
This study aims to determine if there is a link between cow's milk allergy in infants and regulatory T cells dysfunction that should be transient in infant acquiring oral tolerance after 12 month avoiding food and persistent in others.

Cow's milk allergy is evaluated by basophils activation test, T cells activation test, specific humoral response (IgA, IgE, IgG) in allergic infants before and after 12 month avoiding food, before and after low dose milk exposure, before and after oral challenge.

Number and function of regulatory T cells and microflora composition are measured at the same time.

Allergic infants are compared to age matched control group.

ELIGIBILITY:
Inclusion Criteria:

male or female, age before 6 month, cow's milk allergy with positive prick or patch test for cow's milk

Control group: male or female, age before 6 month or within 12 and 18 month, eating cow's milk every day

Exclusion Criteria:

immunodeficiency syndrome, lactose intolerance Control group: other food allergy, atopic dermatitis.

Ages: 1 Month to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Alain LACHAUX, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Alain Lachaux, Lyon, France